CLINICAL TRIAL: NCT05936073
Title: DELTA DESCRIBE: the French Collaborative Project
Acronym: DELTADESCRIBE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: 87RI21_0068
Record Dates: First submitted 2023-06-27; First posted 2023-07-07 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hepatitis D
Keywords: HBs Ag; Delta hepatitis; Screening; Reflex testing
MeSH Terms: conditions — Hepatitis D; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Patients co-infected HBV/HDV — Step 1: collection of SNDS data from 2016 to 2020 Snapshot of the prescription of the Delta tests and the tests usually prescribed simultaneously (HBV but also HIV and HCV) in one year. The investigator will collect the number of tests performed once for a given patient: anti-HDV, HDV RNA, HBsAg, anti-HCV, anti-HIV, and for each test, the description of the profile and the geographical distribution of prescribers in the metropolitan area; the description of age and sex of the patients screened. Step 2: collection of anti-HDV and RNA tests performed in French private and Public laboratories over the year 2019 Anti-HDV and HDV RNA are subcontracted by most private laboratories to two specialized biology companies. Number of HDV tests prescribed, technique used, number of positive tests and name of the requesting laboratory will be collected. The investigator will then go back to the prescriber of the positive tests, identify the patient, his epidemiological profile and his medical care.

SUMMARY:
Our global objective is to draw up a photograph of HDV patients over one year in metropolitan France and identify the barriers of screening and care. The investigator suspects a mismatch between HBV and HDV screening, the first step for specialized care pathway in metropolitan France.

DETAILED DESCRIPTION:
Hepatitis Delta virus (HDV) infection is a significant public health disease causing up to 18% of cirrhosis and 20% of hepatocellular carcinoma (HCC) and new therapeutic options are now available. In France, very few epidemiological studies, mainly focused on specific pre-selected hospital populations, are available. There is a crucial need for data in terms of Delta knowledge, suitability of screening, type of prescribers and treatment access. The investigator proposes a retrospective study in order to describe the number of HDV tests (anti-HDV and HDV RNA) performed in metropolitan France and compare it to the potentially expected one, estimated from the number of HBV screening tests performed in one year, from 2016 to 2020. The investigator will also evaluate the number of HCV and HIV screening tests prescribed over the same period and the HDV PCR techniques used. This study will be based on one hand on data from the French Health insurance (first step) and on the other hand on data from private and hospital laboratories (second step). The second step will allow to identify the prescriber of the Delta tests and the HDV positive patients and precise their profile and their medical care. After an initial analysis of the results, The investigator will propose solutions to the barriers encountered and adapted to the identified targets.

ELIGIBILITY:
Inclusion Criteria:

* >18 years at the second step
* HDV RNA positive patients identified at the second step
* Patients non opposed to the collection of their data

Exclusion Criteria:

* Opposition expressed by the patients for the collection of their data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients (>18 years) chronically infected by HBV and HDV (RNA HDV positive) at the second step
Sampling Method: Non-Probability Sample
Enrollment: 734 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-06-22 (Estimated); Study Completion 2025-06-22 (Estimated)

PRIMARY OUTCOMES:
Number of anti-HDV and HDV RNA tests performed from 2016 to 2020 in metropolitan France | 12 months
  - Number of anti-HDV and HDV RNA tests performed from 2016 to 2020 in metropolitan France according to the French Health insurance database.(SNDS)
Number of anti-HDV and HDV RNA tests expected | 12 months
  - Number of anti-HDV and HDV RNA tests expected over the same period (calculated from the estimate of the positivity of HBsAg tests prescribed in France)

SECONDARY OUTCOMES:
Number of anti-HCV, anti-HIV and HBs Ag tests performed in metropolitan France from 2016 to 2020 | 12 months
  Number of anti-HCV, anti-HIV and HBs Ag performed in France from 2016 to 2020 (SNDS data).
Age, sex, residence department and profile of prescribers of patients receiving HDV, HBV, HIV and HCV tests | 12 months
  Global epidemiological characteristics (age, sex, residence department), of patients receiving HDV, HBV, HIV and HCV tests on the 2016-2020 period, with the profile of prescribers. (SNDS data).
Number of anti-HDV and HDV RNA tests performed in 2019 by the laboratories in metropolitan France | 12 months
  Number and result of anti-HDV and HDV RNA tests performed in 2019 (Private and Public laboratories data
Age, sex, profile of the prescribers of HDV RNA positive patients identified by the laboratories in 2019 | 12 months
  Age, sex, profile of the prescribers, treatment modalities (if available) of HDV RNA positive patients identified at the second step (Private and Public laboratories data)
Rate of use of the different HDV PCR techniques by the laboratories in 2019 | 12 months
  HDV PCR techniques used (Private and Public laboratories data)

CONTACTS AND LOCATIONS:
Overall Officials: Véronique Loustaud-Ratti, Pr, Principal Investigator — University Hospital, Limoges
Locations (1):
- Chu Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No